CLINICAL TRIAL: NCT00323687
Title: Switch to a Completely ONce Daily Regimen Containing Emtricitabine/Tenofovir - Fixed Dose Combination Plus Third QD Partner: "SONETT"
Brief Title: SONETT: Switch Study to Once Daily HIV Treatment Regimen With Truvada
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Thomas Mertenskoetter, Gilead Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-DE-164-0106
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 Infection
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Truvada — 300mg / 200 mg QD tenofovir DF and Emtricitabine Fixed Dose Combination (FDC) Tablet (oral)

SUMMARY:
There is an unmet medical need for potent ART regimens that make adherence to treatment even easier due to QD dosing, offer a good tolerability profile and fit into the daily life of patients.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (over 18 years of age) of any ethnic group without restricted legal competence and who are capable of following the study instructions HIV-1 infection documented by confirmed positive HIV-1 antibody test and/or positive PCR for HIV-1 RNA Stable (no interruption or change of regimen in last 3 months) AZT-and 3TC-containing regimen > 3 months No documented prior virologic failure (virological failure defined as 2 consecutive measurements 4 weeks apart with viral load of HIV-RNA > 400 copies/mL while on ART) CD4+ counts > 50 cells/µL Viral load < 50 copies/mL Karnofsky performance status ≥ 80% For women with childbearing potential, negative urine pregnancy test at Screening visit

Exclusion Criteria:

Serum phosphate level < 0.65 mmol/L Documented active opportunistic infections Subjects with previously documented K65R, 69S mutations or 3 or more thymidine analogue mutations Documented active malignant disease (excluding Kaposi sarcoma limited to the skin) Female of childbearing potential not willing to use a barrier method of contraception during heterosexual intercourse during the duration of study Women who are pregnant or breast feeding Known history of drug, medication or alcohol abuse within the last 12 months preceding the study Simultaneous participation in another study with an investigational drug or within less than one month prior to this study Inability or not willing to meet the requirements of the protocol History of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator Limited mental capacity to the extent that he/she cannot provide informed consent or information regarding adverse events of the study medication Renal disease (creatinine clearance < 50 ml/min according to Cockroft_Gault formula) or severe hepatic, respiratory or cardiovascular disease Patients who have previously been enrolled into this study Contraindication for one of the study substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA < 400 and with HIV RNA < 50 copies/mL at Week 48 | Week 48

SECONDARY OUTCOMES:
Proportion of patients with HIV RNA < 400 and with HIV RNA < 50 copies/mL at Week 24 | 24 weeks
Time to failure or ART discontinuation. Virological failure is defined as 2 consecutive measurements 4 weeks apart with viral load of HIV-RNA > 400 copies/mL | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mertenskoetter, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences GmbH, Martinsried, Germany

REFERENCES:
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-DE-164-0106_synopsis.pdf